CLINICAL TRIAL: NCT06145126
Title: Effects of Glucocortioids in Human Skeletal Muscle, Adipose Tissue and Skin
Acronym: FUSION
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: FUSION
Record Dates: First submitted 2023-10-09; First posted 2023-11-22 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-10

CONDITIONS: Glucocorticoids Toxicity; Iatrogenic Effect
MeSH Terms: interventions — Prednisolone

STUDY DESIGN:
Intervention Model Description: Placebo-controlled, randomized, crossover
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Start pred/End placebo (Other): Both arms will receive both placebo and prednisone
  Interventions: Other: Prednisolone; Other: Placebo
- Start placebo/End pred (Other): Both arms will receive both placebo and prednisone
  Interventions: Other: Prednisolone; Other: Placebo

INTERVENTIONS:
Other: Prednisolone — Predisolone is used as a tool to elicit a physiological response (toolbox trial) and not as a pharmaceutical agent/treatment.
Other: Placebo — Placebo to predinisolon

SUMMARY:
BACKGROUND: A notorious and dreaded adverse effect of glucocorticoids (GC) is redistribution of muscle and fat mass towards muscle wasting and visceral obesity. Fibroadipogenic progenitors (FAPs) are hypothesized to mediate this process.

AIM: Utilizing human data, the investigators study the effects of GC exposure on skeletal muscle structure and function, adipose tissue and skin in healthy older subjects.

METHODS: FAPs will be analyzed in biopsies from skeletal muscles, adipose tissue and skin and further characterized using scRNA-sequencing and Fluorescence-Activated Cell Sorting. Body composition including muscle mass (DXA scan), muscle strength, spontaneous physical activity and glucose homeostasis are recorded.

PERSPECTIVES: The investigators combine translational research with multidisciplinary and international collaboration to elucidate the pathophysiology of GC excess, which is of significant clinical interest since 3% of the Danish population receive GC treatment.

DETAILED DESCRIPTION:
Design: randomized, double blind, placebo-controlled trial. The aim is to study the effect of short-term GC exposure on skeletal muscle, skin , adipose tissue in 12 healthy adults above the age of 50 years. This age group is close to that of patients receiving short-term, high dose anti-inflammatory prednisolone treatment and thus provides a bridge between a clinically observered problem. The participants will be randomized to receive either prednisolone (37,5mg/d) or placebo treatment for five consecutive days. In addition to muscle, skin, and adipose tissue biopsies and body composition measurement (DXA), each participant will undergo the following measurements before and after the intervention: spontaneous physical activity (actigraphy), ambulatory 24-hour blood pressure, continuous glucose monitoring (CGM), pulse wave velocity (PWV), and muscle strength. Each participant is studied before and after the 5-day treatment period.

Outcomes:

* FAPs expression in skeletal muscle and adipose tissue:

  * Fluorescence Activated Cell Sorting (FACS) mediated quantification, isolation and transcriptomic profiling at population and single-cell level of FAPs, and immunological cells
  * Time-to-first division of isolation FAPs
  * In vitro fibro- and adipogenic differentiation of FAPs
  * Single cell transcriptome analysis (scRNA-seq) to profile cell types in a hypothesis-generating perspective.
* Functional outcomes: Muscle mass and strength (DXA scan and isometric quadriceps strength) and spontaneous physical activity (actigraphy)
* Metabolic outcomes: circadian blood glucose and blood pressure, and basal insulin sensitivity.

ELIGIBILITY:
Inclusion Criteria:

* Written and oral consent prior to study beginning
* Age of or above 50 years
* Healthy (uncomplicated hypertension and hypercholesteroleamia is accepted)
* BMI of or below 35

Exclusion Criteria:

* Consumption of glucocorticoid pharmaceuticals (inhalation steroids, intra-articular or intra-muscular injections, steroid creme group IV-V used in the genital area). Allowed pharmaceuticals: ocular drops, nasal sprays/drops, steroid creme group I-III, steroid creme group IV-V used in non-genital areas
* Alcohol consumption of more than 21 units per week
* Consumption of strong CYP3A4 inhibitors/inducers
* Serious comorbidity (heart, liver, or kidney failure, as well as cooncurrent cancer/chemotherapy treatment)
* High daily activity level (more than 30min per day or more than 2 organized workouts per week)

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2024-08 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
FAPs expression in skeletal muscle, adipose tissue, and skin | 2 Years
  Single cell transcriptome analysis (scRNA-seq) to profile cell types in a hypothesis-generating perspective.

SECONDARY OUTCOMES:
Dual X-ray scan (DXA) | 2 Years
  Bodycomposition (grams)
Metabolic outcomes - Circadian blood glucose | Years
  Blood monitoring using Dexcom censor (unit: mmol/L)
Dynamometer | 2 Years
  Isometric muscle contraction (power)
24h blood pressure | 2 Years
  Systolic and diastolic (mmHg)
Basal insulin sensitivity. | 2 Years
  Blood samples (pmol/L)
Activity level | 2 Years
  Spontanous activity level using a wrist ban monitor (ActiGraph)